CLINICAL TRIAL: NCT02632110
Title: A Phase 2 Study of the Effect of Microneedle Lesion Preparation, Incubation Time and Light Power Density on Photodynamic Therapy With Levulan Kerastick (Aminolevulinic Acid HCl) for Topical Solution, 20% + Blue Light for the Field Treatment of Actinic Keratoses on the Face
Brief Title: Microneedle Lesion Preparation Prior to Aminolevulinic Acid Photodynamic Therapy (ALA-PDT) for AK on Face
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP0112
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-12

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid; Solutions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- ALA 25 min 10 Milliwatts (mW) (Experimental): ALA-PDT, 25 min incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  Interventions: Drug: ALA; Device: IBL 10 mW
- MN + ALA 25 min 10 mW (Experimental): Microneedle lesion preparation prior to ALA-PDT, 25 min incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  Interventions: Drug: ALA; Device: IBL 10 mW; Procedure: Microneedle lesion preparation
- ALA 25 min 20 mW (Experimental): ALA-PDT, 25 min incubation period, 20 mW/cm2 power density for 8 min 20 second light treatment.
  Interventions: Drug: ALA; Device: IBL 20 mW
- MN + ALA 25 min 20 mW (Experimental): Microneedle lesion preparation prior to ALA-PDT, 25 min incubation period, 20 mW/cm2 power density for 8 min 20 second light treatment.
  Interventions: Drug: ALA; Procedure: Microneedle lesion preparation; Device: IBL 20 mW
- ALA 60 min 10 mW (Experimental): ALA-PDT, 60 min incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  Interventions: Drug: ALA; Device: IBL 10 mW
- MN + ALA 60 min 10 mW (Experimental): Microneedle lesion preparation prior to ALA-PDT, 60 min incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  Interventions: Drug: ALA; Device: IBL 10 mW; Procedure: Microneedle lesion preparation
- ALA 60 min 20 mW (Experimental): ALA-PDT, 60 min incubation period, 20 mW/cm2 power density for 8 min 20 second light treatment.
  Interventions: Drug: ALA; Device: IBL 20 mW
- MN + ALA 60 min 20 mW (Experimental): Microneedle lesion preparation prior to ALA-PDT, 60 min incubation period, 20 mW/cm2 power density for 8 min 20 second light treatment.
  Interventions: Drug: ALA; Procedure: Microneedle lesion preparation; Device: IBL 20 mW
- VEH (Placebo Comparator): Vehicle (VEH) PDT, 60 minute incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  Interventions: Drug: Topical Solution Vehicle; Device: IBL 10 mW
- MN + VEH (Placebo Comparator): Microneedle lesion preparation prior to Vehicle PDT, 60 minute incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  Interventions: Drug: Topical Solution Vehicle; Device: IBL 10 mW; Procedure: Microneedle lesion preparation

INTERVENTIONS:
Drug: ALA — 20% ALA applied to face prior to light treatment
  Other Names: Levulan Kerastick; Aminolevulinic acid
  Arms: ALA 25 min 10 Milliwatts (mW); ALA 25 min 20 mW; ALA 60 min 10 mW; ALA 60 min 20 mW; MN + ALA 25 min 10 mW; MN + ALA 25 min 20 mW; MN + ALA 60 min 10 mW; MN + ALA 60 min 20 mW
Drug: Topical Solution Vehicle — Levulan Kerastick containing vehicle ingredients only. Vehicle solution applied to face prior to light treatment
  Arms: MN + VEH; VEH
Device: IBL 10 mW — 10 J/cm2 blue light delivered at 10 mW/cm2 for 16 minutes 40 seconds
  Other Names: Investigational Blue Light (IBL)
  Arms: ALA 25 min 10 Milliwatts (mW); ALA 60 min 10 mW; MN + ALA 25 min 10 mW; MN + ALA 60 min 10 mW; MN + VEH; VEH
Procedure: Microneedle lesion preparation — Microneedling of all visible/palpable AK lesions prior to solution application.
  Arms: MN + ALA 25 min 10 mW; MN + ALA 25 min 20 mW; MN + ALA 60 min 10 mW; MN + ALA 60 min 20 mW; MN + VEH
Device: IBL 20 mW — 10 J/cm2 blue light delivered at 20 mW/cm2 for 8 minutes 20 seconds
  Other Names: Investigational Blue Light
  Arms: ALA 25 min 20 mW; ALA 60 min 20 mW; MN + ALA 25 min 20 mW; MN + ALA 60 min 20 mW

SUMMARY:
The purpose of this study is to determine the viability of microneedle lesion preparation (MN) to enhance treatment benefit when performed prior to ALA PDT to an actinic keratosis (AK) field on the face.

ELIGIBILITY:
Inclusion Criteria:

* Four to eight AKs on the face

Exclusion Criteria:

* Pregnancy
* history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins or photodermatosis
* lesions suspicious for skin cancer (skin cancer not ruled out by biopsy) or untreated skin cancers within the Treatment Area
* skin pathology or condition which could interfere with the evaluation of the test product or requires the use of interfering topical or systemic therapy
* Subject is immunosuppressed
* currently enrolled in an investigational drug or device study
* has received an investigational drug or been treated with an investigational device within 30 days prior to the initiation of treatment
* known sensitivity to one or more of the vehicle components (ethyl alcohol, isopropyl alcohol, laureth 4, polyethylene glycol)
* has an active herpes simplex infection OR a history of 2 or more outbreaks within the past 12 months, on the face
* use of the following topical preparations on the extremity to be treated:

  * Keratolytics including urea (greater than 5%), alpha hydroxyacids [e.g.glycolic acid, lactic acid, etc. greater than 5%], salicylic acid (greater than 2%) within 2 days
  * Curettage or Cryotherapy within 2 weeks of initiation of treatment
  * Retinoids, including tazarotene, adapalene, tretinoin, within 4 weeks
  * Microdermabrasion, laser ablative treatments, ALA-PDT, chemical peels, 5 fluorouracil, diclofenac, ingenol mebutate, imiquimod or other topical treatments for AK within 8 weeks
* use of systemic retinoid therapy within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09-12 (Actual); Study Completion 2016-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Marcus, MD, PhD, Study Director — DUSA Pharmaceuticals, Inc.
Locations (8):
- United States (8):
  - UCSD Dermatology, San Diego, California
  - Therapeutics Clinical Research, San Diego, California
  - MOORE Clinical Research, Inc, Brandon, Florida
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Shideler Clinical Research Center, Carmel, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Virginia Clinical Research, Inc., Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: AK Fields
Groups:
- MN + ALA 25 Min 10 mW: Microneedle lesion preparation prior to ALA-PDT, 25 min incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  ALA: 20% ALA applied to face prior to light treatment
  IBL 10 mW: 10 J/cm2 blue light delivered at 10mW/cm2 for 16 minutes 40 seconds
  Microneedle lesion preparation: Microneedling of all visible/palpable AK lesions prior to solution application
- ALA 25 Min 10 mW: Aminolevulinic acid photodynamic therapy (ALA-PDT), 25 min incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  ALA: 20% ALA applied to face prior to light treatment
  Microneedle (MN): one actinic keratosis (AK) Field (1/2 face) on each subject randomized to microneedle lesion preparation prior to ALA application.
  Investigational Blue Light (IBL) 10 mW: 10 J/cm2 blue light delivered at 10mW/cm2 for 16 minutes 40 seconds
- MN + ALA 25 Min 20 mW: Microneedle lesion preparation prior to ALA-PDT, 25 min incubation period, 20 mW/cm2 power density for 8 min 20 second light treatment.
  ALA: 20% ALA applied to face prior to light treatment
  Microneedle lesion preparation: Microneedling of all visible/palpable AK lesions prior to solution application.
  IBL 20 mW: 10 J/cm2 blue light delivered at 20mW/cm2 for 8 minutes 20 seconds
- ALA 25 Min 20 mW: ALA-PDT, 25 min incubation period, 20 mW/cm2 power density for 8 min 20 second light treatment.
  ALA: 20% ALA applied to face prior to light treatment
  MN: one AK Field (1/2 face) on each subject randomized to microneedle lesion preparation prior to ALA application.
  IBL 20 mW: 10 J/cm2 blue light delivered at 20mW/cm2 for 8 minutes 20 seconds
- MN + ALA 60 Min 10mW: Microneedle lesion preparation prior to ALA-PDT, 60 min incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  ALA: 20% ALA applied to face prior to light treatment
  IBL 10 mW: 10 J/cm2 blue light delivered at 10mW/cm2 for 16 minutes 40 seconds
  Microneedle lesion preparation: Microneedling of all visible/palpable AK lesions prior to solution application.
- ALA 60 Min 10 mW: ALA-PDT, 60 min incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  ALA: 20% ALA applied to face prior to light treatment
  MN: one AK Field (1/2 face) on each subject randomized to microneedle lesion preparation prior to ALA application.
  IBL 10 mW: 10 J/cm2 blue light delivered at 10mW/cm2 for 16 minutes 40 seconds
- MN + ALA 60 Min 20 mW: Microneedle lesion preparation prior to ALA-PDT, 60 min incubation period, 20 mW/cm2 power density for 8 min 20 second light treatment.
  ALA: 20% ALA applied to face prior to light treatment
  Microneedle lesion preparation: Microneedling of all visible/palpable AK lesions prior to solution application.
  IBL 20 mW: 10 J/cm2 blue light delivered at 20mW/cm2 for 8 minutes 20 seconds
- ALA 60 Min 20 mW: ALA-PDT, 60 min incubation period, 20 mW/cm2 power density for 8 min 20 second light treatment.
  ALA: 20% ALA applied to face prior to light treatment
  MN: one AK Field (1/2 face) on each subject randomized to microneedle lesion preparation prior to ALA application.
  IBL 20 mW: 10 J/cm2 blue light delivered at 20mW/cm2 for 8 minutes 20 seconds
- MN + VEH 60 Min 10 mW: Microneedle lesion preparation prior to Vehicle PDT, 60 minute incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  Topical Solution Vehicle: Levulan Kerastick containing vehicle ingredients only. Vehicle solution applied to face prior to light treatment
  IBL 10 mW: 10 J/cm2 blue light delivered at 10mW/cm2 for 16 minutes 40 seconds
  Microneedle lesion preparation: Microneedling of all visible/palpable AK lesions prior to solution application
- VEH 60 Min 10 mW: Vehicle (VEH) PDT, 60 minute incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  MN: one AK Field (1/2 face) on each subject randomized to microneedle lesion preparation prior to VEH application.
  Topical Solution Vehicle: Levulan Kerastick containing vehicle ingredients only. Vehicle solution applied to face prior to light treatment
  IBL 10 mW: 10 J/cm2 blue light delivered at 10mW/cm2 for 16 minutes 40 seconds
Period: Overall Study
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH 60 Min 10 mW | VEH 60 Min 10 mW
Started | 25; 25 AK Fields | 25; 25 AK Fields | 27; 27 AK Fields | 27; 27 AK Fields | 29; 29 AK Fields | 29; 29 AK Fields | 26; 26 AK Fields | 26; 26 AK Fields | 30; 30 AK Fields | 30; 30 AK Fields
Completed | 24; 24 AK Fields | 24; 24 AK Fields | 27; 27 AK Fields | 27; 27 AK Fields | 28; 28 AK Fields | 28; 28 AK Fields | 23; 23 AK Fields | 23; 23 AK Fields | 29; 29 AK Fields | 29; 29 AK Fields
Not Completed | 1; 1 AK Fields | 1; 1 AK Fields | 0; 0 AK Fields | 0; 0 AK Fields | 1; 1 AK Fields | 1; 1 AK Fields | 3; 3 AK Fields | 3; 3 AK Fields | 1; 1 AK Fields | 1; 1 AK Fields
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- ALA 25 Min 10 mW: ALA-PDT, 25 min incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  ALA: 20% ALA applied to face prior to light treatment
  MN: one AK Field (1/2 face) on each subject randomized to microneedle lesion preparation prior to ALA application.
  IBL 10 mW: 10 J/cm2 blue light delivered at 10mW/cm2 for 16 minutes 40 seconds
- VEH 60 Min 10 mW: Vehicle PDT, 60 minute incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  MN: one AK Field (1/2 face) on each subject randomized to microneedle lesion preparation prior to VEH application.
  Topical Solution Vehicle: Levulan Kerastick containing vehicle ingredients only. Vehicle solution applied to face prior to light treatment
  IBL 10 mW: 10 J/cm2 blue light delivered at 10mW/cm2 for 16 minutes 40 seconds
- Total: Total of all reporting groups
Arm/Group | ALA 25 Min 10 mW | ALA 25 Min 20 mW | ALA 60 Min 10 mW | ALA 60 Min 20 mW | VEH 60 Min 10 mW | Total
Number analyzed (Participants) | 25 | 27 | 29 | 26 | 30 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (10) | 64 (8) | 67 (8) | 66 (9) | 64 (10) | 65 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 5 | 6 | 3 | 29
  Male | 17 | 20 | 24 | 20 | 27 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 25 | 27 | 28 | 26 | 30 | 136
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 25 | 27 | 29 | 26 | 30 | 137
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Skin Type staging:
  Skin Type I - Burns easily, never tans Skin Type II - Burns easily, tans minimally Skin Type III - Burns moderately, tans gradually Skin Type IV - Burns minimally, tans well
  Participants
    Type I - Burns easily, never tans | 3 | 2 | 2 | 0 | 0 | 7
    Type II - Burns easily, tans minimally | 10 | 12 | 19 | 14 | 21 | 76
    Type III - Burns moderately, tans gradually | 12 | 11 | 6 | 10 | 9 | 48
    Type IV - Burns minimally, tans well | 0 | 2 | 2 | 2 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Complete Clearance Rate
Description: Number of AK Fields with 0 lesions
Time Frame: Week 12
Population: Split-face study
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Groups:
- ALA 25 Min 10 mW: ALA-PDT, 25 min incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  ALA: 20% ALA applied to face prior to light treatment
  IBL 10 mW: 10 J/cm2 blue light delivered at 10mW/cm2 for 16 minutes 40 seconds
- ALA 25 Min 20 mW: ALA-PDT, 25 min incubation period, 20 mW/cm2 power density for 8 min 20 second light treatment.
  ALA: 20% ALA applied to face prior to light treatment
  IBL 20 mW: 10 J/cm2 blue light delivered at 20mW/cm2 for 8 minutes 20 seconds
- ALA 60 Min 10 mW: ALA-PDT, 60 min incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  ALA: 20% ALA applied to face prior to light treatment
  IBL 10 mW: 10 J/cm2 blue light delivered at 10mW/cm2 for 16 minutes 40 seconds
- ALA 60 Min 20 mW: ALA-PDT, 60 min incubation period, 20 mW/cm2 power density for 8 min 20 second light treatment.
  ALA: 20% ALA applied to face prior to light treatment
  IBL 20 mW: 10 J/cm2 blue light delivered at 20mW/cm2 for 8 minutes 20 seconds
- MN + VEH: Microneedle lesion preparation prior to Vehicle PDT, 60 minute incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  Topical Solution Vehicle: Levulan Kerastick containing vehicle ingredients only. Vehicle solution applied to face prior to light treatment
  IBL 10 mW: 10 J/cm2 blue light delivered at 10mW/cm2 for 16 minutes 40 seconds
  Microneedle lesion preparation: Microneedling of all visible/palpable AK lesions prior to solution application.
- VEH PDT: Vehicle PDT, 60 minute incubation period, 10 mW/cm2 power density for 16 min 40 second light treatment.
  Topical Solution Vehicle: Levulan Kerastick containing vehicle ingredients only. Vehicle solution applied to face prior to light treatment
  IBL 10 mW: 10 J/cm2 blue light delivered at 10mW/cm2 for 16 minutes 40 seconds
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 28 | 28 | 23 | 23 | 29 | 29
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 28 | 28 | 23 | 23 | 29 | 29
AK Fields | 16 | 15 | 10 | 12 | 19 | 15 | 18 | 18 | 4 | 4

2. Secondary Outcome: Complete Clearance Rate
Description: Number of AK Fields with 0 Lesions
Time Frame: Week 8
Population: split-face. Week 8 number of participants and units analyzed is based on observed data at that Visit. Number of subjects at Week 8 may differ from number of subjects completing study as noted in participant flow.
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 27 | 27 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 27 | 27 | 25 | 25 | 30 | 30
AK Fields | 5 | 7 | 7 | 7 | 13 | 11 | 8 | 9 | 4 | 2

3. Secondary Outcome: Subject Satisfaction Score
Description: Subject satisfaction score
  1. = Excellent (very satisfied)
  2. = Good (moderately satisfied)
  3. = Fair (slightly satisfied)
  4. = Poor (not satisfied at all)
Time Frame: Week 12
Population: split-face.
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 26 | 26 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 26 | 26 | 30 | 30
AK Fields
  Excellent (very satisfied) | 15 | 13 | 21 | 21 | 18 | 18 | 15 | 14 | 8 | 8
  Good (moderately satisfied) | 8 | 10 | 5 | 5 | 10 | 9 | 7 | 8 | 3 | 3
  Fair (slightly satisfied) | 1 | 1 | 1 | 1 | 0 | 1 | 4 | 4 | 7 | 7
  Poor (not satisfied) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 12

4. Secondary Outcome: Baseline AKCR
Description: AK clearance rate (AKCR) for only those lesions present at Baseline
Time Frame: Baseline and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage cleared
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 27 | 27 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 27 | 27 | 25 | 25 | 30 | 30
percentage cleared | 74.5 (24.14) | 72.3 (30.15) | 75.0 (27.03) | 69.6 (31.4) | 85.4 (22.26) | 83.4 (22.63) | 86.1 (15.59) | 80.6 (22.61) | 40.6 (35.66) | 34.4 (36.66)

5. Secondary Outcome: Baseline AKCR
Description: AK clearance rate for only those lesions present at Baseline
Time Frame: Baseline and Week 12
Population: split-face
Measure: Mean (Standard Deviation); unit: percentage cleared
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 28 | 28 | 23 | 23 | 29 | 29
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 28 | 28 | 23 | 23 | 29 | 29
percentage cleared | 92.2 (16.28) | 89.2 (19.96) | 82.3 (22.32) | 86.7 (16.44) | 93.2 (13.04) | 95.1 (10.4) | 96.3 (7.49) | 94.8 (13.34) | 40.9 (37.24) | 43.1 (40.42)

6. Secondary Outcome: Percent Change
Description: Percent change in the total AK number as compared with Baseline
Time Frame: Baseline and Week 8
Population: split face. Week 8 number of participants and units analyzed is based on observed data at that Visit. Number of subjects at Week 8 may differ from number of subjects completing study as noted in participant flow.
Measure: Mean (Standard Deviation); unit: percent change
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 27 | 27 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 27 | 27 | 25 | 25 | 30 | 30
percent change | -65.9 (28.4) | -68.6 (30.99) | -64.7 (32.32) | -63.4 (36.04) | -72.9 (29.58) | -69.6 (34.46) | -79.4 (17.3) | -74.2 (28.56) | -27.9 (47.29) | -13.8 (49.02)

7. Secondary Outcome: Percent Change
Description: Percent change in the total AK number as compared with Baseline
Time Frame: Baseline and Week 12
Population: split-face
Measure: Mean (Standard Deviation); unit: percent change
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 28 | 28 | 23 | 23 | 29 | 29
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 28 | 28 | 23 | 23 | 29 | 29
percent change | -87.0 (22.52) | -87.3 (20.45) | -75.0 (32.35) | -80.0 (25.1) | -88.9 (21.36) | -87.4 (17.47) | -95.5 (10.16) | -92.6 (19.08) | -26.0 (50.29) | -18.5 (54.77)

8. Other Pre Specified Outcome: Hyperpigmentation
Description: HYPERPIGMENTATION SCALE Grade 0 = No hyperpigmentation Grade 1 = Light hyperpigmentation involving small areas Grade 2 = Moderate hyperpigmentation involving small areas; light hyperpigmentation involving moderate areas Grade 3 = Moderate hyperpigmentation involving moderate sized areas; light hyperpigmentation involving large areas; small areas of marked hyperpigmentation Grade 4 = Marked hyperpigmentation involving moderate or large sized areas
Time Frame: Baseline
Population: split-face
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
AK Fields
  Grade 0 | 12 | 12 | 16 | 16 | 16 | 16 | 13 | 13 | 15 | 15
  Grade 1 | 10 | 11 | 6 | 6 | 11 | 9 | 8 | 8 | 12 | 13
  Grade 2 | 2 | 1 | 5 | 5 | 1 | 3 | 3 | 3 | 1 | 0
  Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
  Grade 4 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1

9. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 8
Time Frame: 24-48 hours after PDT #1
Population: split-face. Number of participants and units analyzed is based on observed data at this visit. Number of subjects with observed data at this visit may differ from number of subjects at baseline or completing study as noted in participant flow.
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
AK Fields
  Grade 0 | 12 | 12 | 15 | 15 | 14 | 15 | 10 | 10 | 15 | 15
  Grade 1 | 11 | 11 | 6 | 7 | 11 | 10 | 11 | 11 | 12 | 13
  Grade 2 | 1 | 1 | 6 | 5 | 2 | 2 | 1 | 2 | 1 | 0
  Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1
  Grade 4 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1

10. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 8
Time Frame: 2 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
AK Fields
  Grade 0 | 11 | 11 | 14 | 14 | 16 | 16 | 12 | 12 | 16 | 15
  Grade 1 | 12 | 12 | 8 | 8 | 9 | 9 | 8 | 8 | 11 | 13
  Grade 2 | 1 | 1 | 5 | 5 | 2 | 2 | 2 | 3 | 2 | 0
  Grade 3 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2
  Grade 4 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0

11. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 8
Time Frame: 8 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 27 | 27 | 24 | 24 | 29 | 29
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 27 | 27 | 24 | 24 | 29 | 29
AK Fields
  Grade 0 | 11 | 11 | 16 | 16 | 16 | 16 | 10 | 10 | 16 | 16
  Grade 1 | 11 | 11 | 6 | 6 | 7 | 8 | 9 | 9 | 10 | 10
  Grade 2 | 1 | 1 | 5 | 5 | 3 | 2 | 3 | 3 | 1 | 1
  Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2
  Grade 4 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0

12. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 8
Time Frame: 12 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 28 | 28 | 24 | 24 | 30 | 30
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 28 | 28 | 24 | 24 | 30 | 30
AK Fields
  Grade 0 | 10 | 10 | 15 | 15 | 19 | 19 | 10 | 10 | 16 | 16
  Grade 1 | 12 | 12 | 7 | 7 | 8 | 8 | 10 | 9 | 10 | 11
  Grade 2 | 1 | 1 | 5 | 5 | 0 | 0 | 1 | 3 | 2 | 1
  Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2
  Grade 4 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0

13. Other Pre Specified Outcome: Hypopigmentation
Description: HYPOPIGMENTATION SCALE Grade 0 = No hypopigmentation Grade 1 = Light hypopigmentation involving small areas Grade 2 = Moderate hypopigmentation involving small areas; light hypopigmentation involving moderate areas Grade 3 = Moderate hypopigmentation involving moderate sized areas; light hypopigmentation involving large areas; small areas of marked hypopigmentation Grade 4 = Marked hypopigmentation involving moderate or large sized areas
Time Frame: Baseline
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
AK Fields
  Grade 0 | 16 | 18 | 20 | 21 | 23 | 24 | 20 | 20 | 25 | 26
  Grade 1 | 8 | 6 | 7 | 6 | 5 | 4 | 5 | 5 | 5 | 4
  Grade 2 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 01 | 1 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 13
Time Frame: 24-48 hours after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
AK Fields
  Grade 0 | 17 | 18 | 20 | 21 | 22 | 23 | 18 | 18 | 26 | 27
  Grade 1 | 7 | 6 | 7 | 6 | 5 | 4 | 5 | 5 | 4 | 3
  Grade 2 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 13
Time Frame: 2 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
AK Fields
  Grade 0 | 15 | 17 | 21 | 22 | 21 | 23 | 16 | 16 | 25 | 26
  Grade 1 | 9 | 7 | 6 | 5 | 7 | 4 | 8 | 8 | 5 | 4
  Grade 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

16. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 13
Time Frame: 8 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 27 | 27 | 24 | 24 | 29 | 29
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 27 | 27 | 24 | 24 | 29 | 29
AK Fields
  Grade 0 | 15 | 17 | 21 | 21 | 18 | 19 | 15 | 15 | 23 | 23
  Grade 1 | 8 | 6 | 6 | 6 | 8 | 7 | 8 | 8 | 6 | 6
  Grade 2 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

17. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 13
Time Frame: 12 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 28 | 28 | 24 | 24 | 30 | 30
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 28 | 28 | 24 | 24 | 30 | 30
AK Fields
  Grade 0 | 16 | 18 | 18 | 20 | 21 | 21 | 16 | 16 | 23 | 22
  Grade 1 | 7 | 5 | 9 | 7 | 7 | 7 | 7 | 7 | 7 | 8
  Grade 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

18. Other Pre Specified Outcome: Erythema
Description: Erythema Scale - Grade 0 = None Grade 1 = Minimal - barely perceptible erythema Grade 2 = Mild - predominantly minimal erythema (pink) in the treated area with or without a few isolated areas of more intense erythema Grade 3 = Moderate - predominantly moderate erythema (red) in the treated area with or without a few isolated areas of intense erythema (bright red) Grade 4 = Severe - predominantly intense erythema (bright red) in the treated area with or without a few isolated areas of very intense (fiery red) erythema
Time Frame: Baseline
Population: split face
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
AK Fields
  Grade 0 | 12 | 12 | 16 | 16 | 17 | 16 | 16 | 15 | 15 | 15
  Grade 1 | 10 | 11 | 8 | 8 | 12 | 12 | 9 | 9 | 12 | 11
  Grade 2 | 2 | 1 | 3 | 3 | 0 | 1 | 1 | 2 | 3 | 4
  Grade 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Other Pre Specified Outcome: Erythema
Description: as for outcome 18
Time Frame: 5 minutes after PDT #1
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 26 | 26 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 26 | 26 | 30 | 30
AK Fields
  Grade 0 | 3 | 4 | 3 | 3 | 2 | 2 | 1 | 1 | 12 | 12
  Grade 1 | 3 | 5 | 9 | 9 | 2 | 4 | 6 | 8 | 7 | 9
  Grade 2 | 15 | 13 | 4 | 7 | 12 | 12 | 9 | 10 | 10 | 8
  Grade 3 | 4 | 3 | 11 | 8 | 12 | 10 | 9 | 5 | 1 | 1
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0

20. Other Pre Specified Outcome: Erythema
Description: as for outcome 18
Time Frame: 24-48 hours after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
AK Fields
  Grade 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 11 | 12
  Grade 1 | 0 | 0 | 1 | 2 | 2 | 3 | 0 | 2 | 9 | 10
  Grade 2 | 11 | 14 | 9 | 14 | 6 | 9 | 10 | 10 | 10 | 8
  Grade 3 | 14 | 10 | 13 | 8 | 17 | 12 | 12 | 9 | 0 | 0
  Grade 4 | 0 | 0 | 3 | 2 | 3 | 4 | 3 | 4 | 0 | 0

21. Other Pre Specified Outcome: Erythema
Description: as for outcome 18
Time Frame: 2 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
AK Fields
  Grade 0 | 9 | 10 | 14 | 14 | 15 | 15 | 12 | 13 | 13 | 13
  Grade 1 | 13 | 11 | 9 | 10 | 9 | 10 | 11 | 9 | 14 | 14
  Grade 2 | 3 | 3 | 4 | 3 | 4 | 3 | 2 | 3 | 3 | 3
  Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Other Pre Specified Outcome: Erythema
Description: as for outcome 18
Time Frame: 8 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 27 | 27 | 24 | 24 | 29 | 29
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 27 | 27 | 24 | 24 | 29 | 29
AK Fields
  Grade 0 | 12 | 12 | 16 | 18 | 18 | 17 | 16 | 15 | 14 | 14
  Grade 1 | 10 | 10 | 9 | 7 | 7 | 8 | 7 | 9 | 10 | 10
  Grade 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 0 | 5 | 5
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Other Pre Specified Outcome: Erythema
Description: as for outcome 18
Time Frame: 12 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 28 | 28 | 24 | 24 | 30 | 30
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 28 | 28 | 24 | 24 | 30 | 30
AK Fields
  Grade 0 | 15 | 14 | 19 | 18 | 20 | 19 | 16 | 17 | 15 | 14
  Grade 1 | 7 | 8 | 7 | 8 | 7 | 8 | 8 | 7 | 8 | 9
  Grade 2 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 7 | 7
  Grade 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Other Pre Specified Outcome: Edema
Description: EDEMA SCALE Grade 0 = None Grade 1 = Minimal - scant, rare edema Grade 2 = Mild - easily seen edema, minimally palpable, involving up to 1/3 of the treatment area Grade 3 = Moderate - easily seen edema and typically palpable, involving between 1/3 to 2/3 of the treatment area Grade 4 = Severe - easily seen edema, indurated in some areas, involving over 2/3 of the treatment area
Time Frame: Baseline
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
AK Fields
  Grade 0 | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
  Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Other Pre Specified Outcome: Edema
Description: as for outcome 24
Time Frame: 5 minutes after PDT #1
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 26 | 26 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 26 | 26 | 30 | 30
AK Fields
  Grade 0 | 20 | 20 | 23 | 23 | 23 | 26 | 22 | 24 | 29 | 28
  Grade 1 | 3 | 4 | 2 | 3 | 5 | 1 | 2 | 1 | 1 | 2
  Grade 2 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Other Pre Specified Outcome: Edema
Description: as for outcome 24
Time Frame: 24-48 hours after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
AK Fields
  Grade 0 | 13 | 18 | 20 | 20 | 17 | 14 | 8 | 13 | 29 | 29
  Grade 1 | 8 | 4 | 3 | 3 | 5 | 9 | 9 | 5 | 0 | 1
  Grade 2 | 3 | 2 | 3 | 3 | 4 | 3 | 6 | 3 | 1 | 0
  Grade 3 | 1 | 1 | 1 | 1 | 2 | 2 | 2 | 3 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

27. Other Pre Specified Outcome: Edema
Description: as for outcome 24
Time Frame: 2 weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
AK Fields
  Grade 0 | 25 | 24 | 25 | 25 | 28 | 28 | 24 | 25 | 30 | 30
  Grade 1 | 0 | 1 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

28. Other Pre Specified Outcome: Edema
Description: as for outcome 24
Time Frame: 8 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 27 | 27 | 24 | 24 | 29 | 29
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 27 | 27 | 24 | 24 | 29 | 29
AK Fields
  Grade 0 | 24 | 24 | 27 | 27 | 27 | 27 | 24 | 24 | 29 | 29
  Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

29. Other Pre Specified Outcome: Edema
Description: as for outcome 24
Time Frame: 12 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 28 | 28 | 24 | 24 | 30 | 30
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 28 | 28 | 24 | 24 | 30 | 30
AK Fields
  Grade 0 | 24 | 24 | 27 | 27 | 28 | 28 | 24 | 24 | 30 | 30
  Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

30. Other Pre Specified Outcome: Stinging/Burning
Description: STINGING AND BURNING SCALE Grade 0 = None Grade 1 = Minimal, barely perceptible -tolerable and little discomfort Grade 2 = Moderate - tolerable, but causes some discomfort Grade 3 = Severe - very uncomfortable or intolerable
Time Frame: Baseline
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
AK Fields
  Grade 0 | 24 | 24 | 27 | 27 | 29 | 29 | 25 | 25 | 29 | 30
  Grade 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

31. Other Pre Specified Outcome: Stinging/Burning
Description: Immediately after PDT, the most intensive, acute perception of Stinging/Burning DURING treatment will be recorded.
  STINGING AND BURNING SCALE Grade 0 = None Grade 1 = Minimal, barely perceptible -tolerable and little discomfort Grade 2 = Moderate - tolerable, but causes some discomfort Grade 3 = Severe - very uncomfortable or intolerable
Time Frame: During PDT #1
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
AK Fields
  Grade 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 21 | 24
  Grade 1 | 9 | 14 | 7 | 16 | 5 | 5 | 5 | 6 | 9 | 6
  Grade 2 | 13 | 9 | 16 | 7 | 15 | 17 | 10 | 12 | 0 | 0
  Grade 3 | 2 | 0 | 3 | 3 | 9 | 7 | 11 | 8 | 0 | 0

32. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 30
Time Frame: 5 minutes after PDT #1
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 26 | 26 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 26 | 26 | 30 | 30
AK Fields
  Grade 0 | 6 | 9 | 7 | 9 | 5 | 5 | 5 | 7 | 28 | 29
  Grade 1 | 16 | 14 | 12 | 13 | 16 | 19 | 9 | 11 | 2 | 1
  Grade 2 | 3 | 2 | 8 | 5 | 7 | 4 | 11 | 7 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

33. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 30
Time Frame: 24-48 Hours after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
AK Fields
  Grade 0 | 9 | 8 | 12 | 13 | 7 | 6 | 8 | 9 | 28 | 28
  Grade 1 | 6 | 14 | 8 | 11 | 15 | 16 | 9 | 10 | 2 | 2
  Grade 2 | 10 | 3 | 6 | 3 | 6 | 6 | 8 | 6 | 0 | 0
  Grade 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

34. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 30
Time Frame: 2 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
AK Fields
  Grade 0 | 24 | 24 | 26 | 26 | 28 | 28 | 25 | 25 | 30 | 30
  Grade 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

35. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 30
Time Frame: 8 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 27 | 27 | 24 | 24 | 29 | 29
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 27 | 27 | 24 | 24 | 29 | 29
AK Fields
  Grade 0 | 24 | 24 | 27 | 27 | 27 | 27 | 23 | 22 | 28 | 29
  Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

36. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 30
Time Frame: 12 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 28 | 28 | 24 | 24 | 30 | 30
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 28 | 28 | 24 | 24 | 30 | 30
AK Fields
  Grade 0 | 24 | 24 | 27 | 26 | 27 | 27 | 24 | 24 | 30 | 30
  Grade 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

37. Other Pre Specified Outcome: Scaling & Dryness
Description: SCALING AND DRYNESS SCALE Grade 0 = None Grade 1 = Minimal - barely perceptible desquamation Grade 2 = Mild - limited areas of fine desquamation in up to 1/3 of the treatment area Grade 3 = Moderate - fine desquamation involving 1/3 to 2/3 of the treatment area or limited areas of coarser scaling Grade 4 = Severe - coarser scaling involving more than 2/3 of the treatment area or limited areas of very coarse scaling
Time Frame: Baseline
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
AK Fields
  Grade 0 | 19 | 19 | 18 | 18 | 16 | 16 | 17 | 17 | 19 | 19
  Grade 1 | 5 | 5 | 7 | 8 | 12 | 10 | 8 | 7 | 8 | 8
  Grade 2 | 1 | 1 | 2 | 0 | 1 | 3 | 1 | 2 | 3 | 3
  Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

38. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 37
Time Frame: 24-48 hours after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
AK Fields
  Grade 0 | 15 | 15 | 16 | 17 | 16 | 17 | 17 | 16 | 20 | 20
  Grade 1 | 7 | 7 | 7 | 7 | 6 | 7 | 3 | 6 | 7 | 8
  Grade 2 | 1 | 2 | 3 | 3 | 4 | 2 | 3 | 2 | 2 | 1
  Grade 3 | 2 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 1
  Grade 4 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

39. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 37
Time Frame: 2 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
AK Fields
  Grade 0 | 16 | 17 | 16 | 16 | 20 | 21 | 20 | 21 | 22 | 23
  Grade 1 | 8 | 7 | 10 | 7 | 5 | 4 | 3 | 1 | 8 | 7
  Grade 2 | 0 | 0 | 1 | 4 | 3 | 3 | 1 | 2 | 0 | 0
  Grade 3 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

40. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 37
Time Frame: 8 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 27 | 27 | 24 | 24 | 29 | 29
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 27 | 27 | 24 | 24 | 29 | 29
AK Fields
  Grade 0 | 19 | 20 | 20 | 21 | 22 | 22 | 18 | 19 | 22 | 22
  Grade 1 | 4 | 3 | 6 | 5 | 3 | 3 | 4 | 3 | 4 | 3
  Grade 2 | 0 | 0 | 1 | 1 | 2 | 2 | 2 | 2 | 2 | 3
  Grade 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

41. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 37
Time Frame: 12 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 28 | 28 | 24 | 24 | 30 | 30
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 28 | 28 | 24 | 24 | 30 | 30
AK Fields
  Grade 0 | 23 | 22 | 23 | 22 | 25 | 24 | 20 | 21 | 23 | 23
  Grade 1 | 0 | 1 | 4 | 5 | 3 | 3 | 3 | 2 | 6 | 6
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
  Grade 3 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

42. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: OOZING/VESICULATION/CRUSTING Grade 0 = None Grade 1 = Minimal - a single area of oozing, vesiculation or crusting 3 mm diameter or less in size Grade 2 = Mild - two to four areas of oozing, vesiculation or crusting 3 mm diameter or less in size OR a single area larger than 3 mm diameter in size Grade 3 = Moderate - more than a single area of oozing, vesiculation or crusting larger than 3 mm diameter in size or more than four areas of 3 mm diameter or less in size Grade 4 = Severe - any degree of oozing, vesiculation or crusting greater than (3) above
Time Frame: Baseline
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 29 | 29 | 26 | 26 | 30 | 30
AK Fields
  Grade 0 | 23 | 24 | 24 | 25 | 29 | 29 | 24 | 24 | 29 | 29
  Grade 1 | 1 | 0 | 2 | 1 | 0 | 0 | 2 | 2 | 0 | 0
  Grade 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

43. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 42
Time Frame: 24-48 hours after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
AK Fields
  Grade 0 | 18 | 20 | 21 | 23 | 24 | 25 | 20 | 19 | 29 | 29
  Grade 1 | 4 | 2 | 3 | 2 | 2 | 1 | 4 | 5 | 0 | 0
  Grade 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1
  Grade 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

44. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 42
Time Frame: 2 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
Number analyzed (AK Fields) | 25 | 25 | 27 | 27 | 28 | 28 | 25 | 25 | 30 | 30
AK Fields
  Grade 0 | 23 | 24 | 25 | 26 | 26 | 27 | 24 | 25 | 28 | 28
  Grade 1 | 1 | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 1 | 1
  Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

45. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 42
Time Frame: 8 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 27 | 27 | 24 | 24 | 29 | 29
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 27 | 27 | 24 | 24 | 29 | 29
AK Fields
  Grade 0 | 23 | 23 | 25 | 25 | 25 | 26 | 23 | 23 | 26 | 26
  Grade 1 | 0 | 0 | 1 | 2 | 2 | 1 | 1 | 1 | 1 | 1
  Grade 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

46. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 42
Time Frame: 12 Weeks after PDT #1
Population: as for outcome 9
Measure: Count of Units; unit: AK Fields
Units Other Than Participants: AK Fields
Arm/Group | MN + ALA 25 Min 10 mW | ALA 25 Min 10 mW | MN + ALA 25 Min 20 mW | ALA 25 Min 20 mW | MN + ALA 60 Min 10mW | ALA 60 Min 10 mW | MN + ALA 60 Min 20 mW | ALA 60 Min 20 mW | MN + VEH | VEH PDT
Number analyzed (Participants) | 24 | 24 | 27 | 27 | 28 | 28 | 24 | 24 | 30 | 30
Number analyzed (AK Fields) | 24 | 24 | 27 | 27 | 28 | 28 | 24 | 24 | 30 | 30
AK Fields
  Grade 0 | 24 | 24 | 27 | 27 | 28 | 28 | 23 | 23 | 29 | 29
  Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: This was a split face study where one AK Field on a subjects was randomized to MN lesion pretreatment and the other AK Field was randomized to no pretreatment, but both Fields received the same drug/light treatment. Local skin tolerability effects were presented separately for +MN and -MN, but AEs were evaluated on a per SUBJECT basis, not on a per FIELD basis.
Arm/Group | ALA 25 Min 10 mW | ALA 25 Min 20 mW | ALA 60 Min 10 mW | ALA 60 Min 20 mW | VEH 60 Min 10 mW
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27 | 0/29 | 0/26 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27 | 0/29 | 1/26 | 0/30
Other Adverse Events (participants affected / at risk) | 1/25 | 1/27 | 4/29 | 7/26 | 2/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALA 25 Min 10 mW (N=25) | ALA 25 Min 20 mW (N=27) | ALA 60 Min 10 mW (N=29) | ALA 60 Min 20 mW (N=26) | VEH 60 Min 10 mW (N=30)
unstable angina (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALA 25 Min 10 mW (N=25) | ALA 25 Min 20 mW (N=27) | ALA 60 Min 10 mW (N=29) | ALA 60 Min 20 mW (N=26) | VEH 60 Min 10 mW (N=30)
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Pain (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
First publication of results will be made by the Sponsor. If publication is not submitted within 12 months after the date of study final report, the PI may publish the results from the site individually, subject to compliance with the other terms of the clinical trial agreement, including a requirement that the PI provide a draft of the publication for the sponsor's review 30 days before submission for publication so that sponsor can review the publication for confidential information